CLINICAL TRIAL: NCT01243164
Title: Efficacy of the Wheelchair Skills Training Program for Improving Confidence With Using a Manual Wheelchair in Younger and Older Able-bodied Adults: A Pilot RCT
Brief Title: Efficacy of Wheelchair Skills Training on Confidence Using a Manual Wheelchair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H10-02385
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Confidence Using a Wheelchair
Keywords: confidence; wheelchair performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wheelchair Skills Training Program (Experimental): A standardized wheelchair skills training program to teach 32 specific wheelchair skills.
  Interventions: Other: Wheelchair Skills Training Program

INTERVENTIONS:
Other: Wheelchair Skills Training Program — The Wheelchair Skills Training Program will be administered in 2, 1 hour sessions.
  Other Names: WSTP

SUMMARY:
Background and Rationale: Mobility impairment is one of the main correlates of decreased levels of participation in daily and social activities. Mobility disability is often remediable through the use of assistive technology, of which the wheelchair is arguably the most widely used and recognizable form. Statistics suggest over 250,000 Canadians use wheelchairs, the majority of whom are older adults.

Mobility impairment often has psychological consequences that may independently restrict functioning and participation. Confidence is one such consequence, and according to Bandura's Social Cognitive Theory, is the belief individuals have in their ability to perform behaviours to achieve desired outcomes. Furthermore, previous findings have accounted for no more than 40% of the variance of factors influencing wheelchair mobility and participation. It is likely that confidence in wheelchair use may account for some of that variance. Recent findings show that approximately 40% of wheelchair users report having low confidence.

Because confidence is client-specific and modifiable, treatment strategies to address low confidence in using a wheelchair may lead to greater participation among older adults.

Purpose: The overall goal of this research project is to evaluate the efficacy of the Wheelchair Skills Training Program on confidence with using a manual wheelchair in a group of non-wheelchair users.

Objectives:

1. Evaluate the efficacy of the Wheelchair Skills Training Program on improving confidence with using a manual wheelchair.
2. Evaluate the efficacy of the Wheelchair Skills Training Program on improving wheelchair performance.
3. Explore the immediate effect of exposure to wheelchair skills (an outcome measure) on confidence using a manual wheelchair.

Hypotheses:

1. Participants who take part in the Wheelchair Skills Training Program will have significant improvements in confidence with using a manual wheelchair compared with those in the control group, as measured by the Wheelchair Use Confidence Scale (WheelCon)
2. Participants who receive the Wheelchair Skills Training Program will have significant improvements in wheelchair performance compared to the control group, as measured by the Wheelchair Skills Test (WST).
3. All participants will have significant improvements in confidence using a manual wheelchair after exposure to wheelchair skills (during baseline assessment).

Research Method: This study will use 2 concurrent Randomized Controlled Trials to evaluate the efficacy of the Wheelchair Skills Training Program in younger and older adults. Trial 1 and Trial 2 will employ different recruitment approaches for targeting younger versus older adults and different inclusion criteria with regard to age of the participants. Otherwise the research design, protocol and procedures will be the same. Upon completion of data collection, the data will be pooled and stratified by age (younger adult, older adult) for analyses.

DETAILED DESCRIPTION:
Background and Rationale:

Mobility impairment is the primary form of reported disability and is also one of the main correlates of decreased levels of participation in daily and social activities, which is an important determinant of quality of life. Mobility disability is often remediable through the use of assistive technology, of which the wheelchair is arguably the most widely used and recognizable form. Statistics suggest over 250,000 Canadians use wheelchairs the majority of whom are older adults.

Sudden health events such as mobility impairment often have psychological consequences that may independently restrict functioning and participation. Confidence is one such consequence, and according to Bandura's Social Cognitive Theory, is the belief individuals have in their ability to perform behaviours to achieve desired outcomes. Furthermore, previous findings have accounted for only 33% and 40% of the variance of factors influencing wheelchair mobility and participation respectively. It is likely that confidence in wheelchair use may account for some of that variance. Confidence in using a wheelchair is an emerging and novel research construct that has the potential for significant impact on healthy and successful aging, and on health services aimed towards the maintenance of functional autonomy among older adults. It is conceptualized as the belief individuals have in their ability to use a wheelchair, and recent findings show that approximately 40% of wheelchair users have low confidence.

Because confidence is client-specific and modifiable, treatment strategies to address low confidence in using a wheelchair may lead to greater mobility and social participation among older adults. Bandura postulates four sources of information to modify confidence: 1) enactive mastery; 2) vicarious learning; 3) verbal persuasion; and 4) physiological/ affective states. Enactive mastery, or experiential learning, is perhaps the most influential source of information. Enactive mastery has been shown to positively alter many forms of confidence including those related to balance, and performance of activities of daily living. In fact, qualitative responses from a community-based study stated that wheelchair users reported increased confidence after completing the Wheelchair Skills Training Program. It is thus plausible that wheelchair skills training may positively influence an older adult's confidence in their ability to use a wheelchair. However, this relationship has not yet been explored.

Purpose: The overall goal of this research project is to evaluate the efficacy of the Wheelchair Skills Training Program on confidence with using a manual wheelchair in younger and older able-bodied adults.

Objectives:

1. Evaluate the efficacy of the Wheelchair Skills Training Program on improving confidence with using a manual wheelchair.
2. Evaluate the efficacy of the Wheelchair Skills Training Program on improving wheelchair performance.
3. Explore the immediate effect of exposure to wheelchair skills on confidence using a manual wheelchair.
4. Evaluate the difference in confidence using a manual wheelchair between younger and older adults.

Hypotheses:

1. Participants who take part in the Wheelchair Skills Training Program will have significant improvements in confidence with using a manual wheelchair compared with those in the control group.
2. Participants who receive the Wheelchair Skills Training Program will have significant improvements in wheelchair performance compared to the control group.
3. Confidence with using a manual wheelchair will improve after exposure to wheelchair skills.
4. Younger adults will have significantly higher confidence using a manual wheelchair compared to older adults.

Research Method: Concurrent Randomized Controlled Trials in a group of younger (Trial 1) and older (Trial 2) adults.

Trial 1- Participants: Undergraduate and graduate, able-bodied students will be recruited through the University of British Columbia using letters of information, posters, and word-of-mouth.

Sample Size: 20 (10 intervention, 10 control)

Trial 2- Participants: Able-bodied community living, older adults Sample Size: 20 (10 intervention, 10 control)

Trial 1 and Trial 2- Design: Parallel group, randomized controlled trial. Procedures: Informed consent will be obtained from interested participants. Demographic information and information about anxiety and depression, cognitive functioning, and risk propensity will be collected. Participants will then be randomly allocated to either a Wheelchair Skills Training Program (WSTP) or a Control group using a table of random numbers.

All participants will complete baseline and follow-up measures for confidence using a manual wheelchair and wheelchair performance. Participants in the intervention group will complete the WSTP, while participants in the control will just receive one phone call or email from the study investigators.

Statistical Analysis: Demographic information, anxiety and depression, cognitive functioning, and risk propensity will be analyzed using descriptive statistics. The change in confidence with using a manual wheelchair between groups (WSTP and Control) will be analyzed using a 2X3X2 repeated measures ANOVA. The change in confidence with using a manual wheelchair between groups (WSTP and Control) will be analyzed using a 2X2X2 repeated measures ANOVA. All data will be analyzed using SPPS Version 15.0, with alpha equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* able-bodied
* 19 years of age or older
* able to propel a manual wheelchair for at least 10 metres

Exclusion Criteria:

* are unable to speak and write in English
* have an upper extremity injury
* use a wheelchair for mobility
* have previously taken part in wheelchair skills training workshops
* have a heart condition that could be worsened by physical activity
* have a physician diagnosis of osteoporosis or osteopenia
* live in residential or long-term care

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Confidence Using a Wheelchair (WheelCon) | 2 weeks
  A 63-item questionnaire to assess confidence using a manual wheelchair

SECONDARY OUTCOMES:
Wheelchair Skills Test (WST) | 2 weeks
  A 32-item performance-based wheelchair obstacle course. The WST assessed the ability to perform a standardized set of wheelchair skills and also assess whether the skills were performed safely
Hospital Anxiety and Depression Scale (HADS) | 2 weeks
  HADS is a 14 item questionnaire to asses anxiety and depression.
Evaluation of Risk scale (EVAR) | 2 weeks
  EVAR is a 24 item questionnaire that assesses propensity of risk taking behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Blusson Spinal Cord Centre, Vancouver, British Columbia
  - GF Strong, Vancouver, British Columbia

REFERENCES:
- See also: Related Info — http://www.wheelchairskillsprogram.ca